CLINICAL TRIAL: NCT01427972
Title: Study of the Safety and Efficacy of LY2623091 in Chronic Kidney Disease Patients
Brief Title: A Study of LY2623091 in Male and Females With Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 14350; I4M-MC-MRAC (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-08-31; First posted 2011-09-02 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-08

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.2 milligrams (mg) LY2623091 (Experimental): Daily by mouth for 21 days. Days 1-20 administered in the fed state. Day 21 administered in the fasted state. Minimum wash-out period of 28 days between dosing in treatment periods
  Interventions: Drug: LY2623091
- 1.5 mg LY2623091 (Experimental): Daily by mouth for 21 days. Days 1-20 administered in the fed state. Day 21 administered in the fasted state. Minimum wash-out period of 28 days between dosing in treatment periods
  Interventions: Drug: LY2623091
- 10 mg LY2623091 (Experimental): Daily by mouth for 21 days. Days 1-20 administered in the fed state. Day 21 administered in the fasted state. Minimum wash-out period of 28 days between dosing in treatment periods
  Interventions: Drug: LY2623091
- 50 mg Eplerenone (Active Comparator): Daily by mouth for 21 days. Days 1-20 administered in the fed state. Day 21 administered in the fasted state. Minimum wash-out period of 28 days between dosing in treatment periods
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: LY2623091 — Administered orally
  Arms: 0.2 milligrams (mg) LY2623091; 1.5 mg LY2623091; 10 mg LY2623091
Drug: Eplerenone — Administered orally
  Arms: 50 mg Eplerenone

SUMMARY:
The purpose of this trial is to investigate the safety and efficacy of LY2623091 in males and females with chronic kidney disease.

DETAILED DESCRIPTION:
This trial consists of 4 treatment arms: 3 LY2623091 dose levels and eplerenone. Each participant will participate in 2 treatment periods, with a minimum wash-out period of 28 days between dosing in the 2 treatment periods. Dosing days will be numbered 1-21 in each of the 2 treatment periods. Participants will receive different treatments in periods 1 and 2. Participants will be housed as inpatients during the days of the controlled diet administration and the oral potassium challenge and until at least 24 hours after its completion (Days -3 to 1; Days 19 to 22, in each treatment period). Otherwise the study will be done on an outpatient basis, with participants returning to the clinic for evaluations during each treatment period (Days 3 or 4, 7, and 14).

ELIGIBILITY:
Inclusion Criteria:

* Men and women of non-childbearing potential as determined by medical history and physical examination

  1. Male participants: Non-vasectomized male participants must agree to use 2 medically accepted methods of contraception with all sexual partners during the study and for 90 days following the final dosing. Medically accepted effective forms of contraception may include condoms with contraceptive foam or having partners use diaphragms with contraceptive jelly or cervical caps with contraceptive jelly
  2. Female participants: Female participants must be of non-childbearing potential due to surgical sterilization (hysterectomy, bilateral oophorectomy or tubal ligation) or menopause. Postmenopausal women should be a minimum of 12 months without a menstrual period. Perimenopausal women who are 6 months without a menstrual period, have a follicle stimulating hormone (FSH) level 23.0-116.3 international unit/liter (IU/L) and are between the ages of 45 and 65 years, inclusive, are also eligible
* Have been diagnosed with Chronic Kidney Disease (CKD) (and including diabetic kidney disease and chronic glomerulonephritis)
* Have an estimated glomerular filtration rate (eGFR) between 30-70 milliliter/minute/1.73 square meters(30-70 ml/min/1.73m²)
* Have been taking an angiotensin converting enzyme (ACE) inhibitor and/or angiotensin II receptor blocker (ARB), for at least 3 months, and at a stable dose for greater than or equal to (≥) 2 months prior to randomization, and agree to continue to take such throughout the duration of the study
* Participants must meet both of the following renal function criteria prior to qualifying for randomization:

  1. Have Screening first morning urine protein/creatinine ratio (PCR) ≥400 milligram/gram (mg/g)
  2. Have stable renal function, in the opinion of the Investigator
* Stable use of blood pressure (BP) medication and acceptable cuff BP, as defined by the following criteria:

  1. While receiving stable dose of an ACE inhibitor and/or ARB
  2. While receiving stable doses of any other applicable BP medication (including diuretic therapy) for ≥3 weeks prior to screening
  3. Have seated cuff systolic BP less than or equal to (≤) 160 millimeters of mercury (mm Hg) and diastolic BP ≤100 mm Hg
* Have serum potassium (K+)≤5.0 milliequivalents/liter (mEq/L) at Screening, and no more that 1 hospitalization due to hyperkalemia within 1 year
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow specific study procedures
* Have venous access sufficient to allow blood sampling
* Have lab values and other safety parameters that are, in the opinion of the investigator, acceptable for participation in the study

Exclusion Criteria:

* Participants who are currently enrolled in, or have discontinued within the last 30 days of the investigational drug from, a clinical trial involving an investigational drug or device or an off-label use of an approved drug (other than the study drug used in this study), or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study. Participants may be enrolled in this study and dosed on day 31 or greater following the last day of previous investigational drug administration
* Have previously completed or withdrawn from this study or any other study investigating LY2623091
* Participants who are taking any diuretic drug and not receiving a stable dose for 3 weeks prior to the screening/qualification visit and through end of treatment
* Participants receiving a renin inhibitor, or an mineralocorticoid receptor (MR) antagonist must have a wash-out period of at least 1 month prior to randomization
* Participants in whom dialysis or renal transplantation is anticipated by their physician within 6 months after the Screening
* Participants with a history of acute kidney injury within 3 months before Screening
* Participants who have or are expected to require systemic immunosuppression therapy within 30 days of Screening(except for inhalant steroids)
* Use of oral or parenteral corticosteroids within 30 days of the Screening
* Participants with a diagnosis of Class three (III) or four (IV) congestive heart failure (CHF) [as defined by the New York Heart Association (NYHA)]
* Participants with evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies; participants with a history of cirrhosis or hepatitis C or are positive for hepatitis C antibody at Screening; participants who are known to be hepatitis B surface antigen-positive or are positive for hepatitis B surface antigen at Screening
* Participants who are unwilling or unable to comply with the use of a data collection device to directly record data from the participants
* Use of a metabolizing enzyme [cytochrome P450 (CYP3A4)] inhibitors or inducers, potassium sparing diuretic drugs (all other diuretic drugs are allowed, potassium supplements or systemic glucocorticoids within 7 days of study enrollment. Intermittent use of nonsteroidal anti-inflammatory drug (NSAIDs) is permitted, except for within 24 hours of critical urine sodium/potassium measures or during the inpatient periods, during which times NSAID use is limited to chronic use only (stable for ≥1 month prior to enrollment). Prostaglandin inhibitors should not be used during the inpatient periods of the study, with above exception of chronic NSAID use
* Have donated blood of more than 500 milliliter (mL) within the last 60 days of screening
* Have an average weekly alcohol intake that exceeds 21 units per week or participants unwilling to stop alcohol intake within 48 hours of entry into study and for the duration of the study [1 unit equal 12 ounces (oz) or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits]
* Evidence of regular use of drugs of abuse
* Consumption of natural licorice and/or natural licorice-containing products and/or regular daily consumption of grapefruit and/or grapefruit juice within 7 days of first dosing and/or anticipated consumption during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sofia, Bulgaria
- South Africa (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloemfontein
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newton Park
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pretoria

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (pts) were randomized to 1 of 4 arms, 3 LY2623091 (LY) and Eplerenone (Epl). Each participated in two 21-day treatment periods with washout period of at least 28 days. Pts who received LY in Period 1 were randomized to a different LY arm or Epl arm in Period 2. Pts who received Epl in Period 1 were randomized to an LY arm in Period 2.
Groups:
- 1.5 mg LY2623091 First Then 10 mg LY2623091: Participants received 1.5 milligram (mg) LY2623091 administered orally, once daily (QD) for 21 days in treatment period 1 followed by a minimum 28-day washout period before receiving 10 mg LY2623091 for 21 days in treatment period 2. On Day 1 through Day 20, participants were in a fed state and on Day 21 participants were in a fasted state.
- 1.5 mg LY2623091 First Then 50 mg Eplerenone: Participants received 1.5 mg LY2623091 administered orally, QD for 21 days in treatment period 1 followed by a minimum 28-day washout period before receiving 50 mg Eplerenone for 21 days in treatment period 2. On Day 1 through Day 20, participants were in a fed state and on Day 21 participants were in a fasted state.
- 1.5 mg LY2623091 First Then 0.2 mg LY2623091: Participants received 1.5 mg LY2623091 administered orally, QD for 21 days in treatment period 1 followed by a minimum 28-day washout period before receiving 0.2 mg LY2623091 for 21 days in treatment period 2. On Day 1 through Day 20, participants were in a fed state and on Day 21 participants were in a fasted state.
- 50mg Eplerenone First Then 0.2 mg LY2623091: Participants received 50 mg Eplerenone administered orally, QD for 21 days in treatment period 1 followed by a minimum 28-day washout period before receiving 0.2 mg LY2623091 for 21 days in treatment period 2. On Day 1 through Day 20, participants were in a fed state and on Day 21 participants were in a fasted state.
- 50mg Eplerenone First Then 1.5 mg LY2623091: Participants received 50 mg Eplerenone administered orally, QD for 21 days in treatment period 1 followed by a minimum 28-day washout period before receiving 1.5 mg LY2623091 for 21 days in treatment period 2. On Day 1 through Day 20, participants were in a fed state and on Day 21 participants were in a fasted state.
- 50mg Eplerenone First Then 10 mg LY2623091: Participants received 50 mg Eplerenone administered orally, QD for 21 days in treatment period 1 followed by a minimum 28-day washout period before receiving 10 mg LY2623091 for 21 days in treatment period 2. On Day 1 through Day 20, participants were in a fed state and on Day 21 participants were in a fasted state.
- 0.2 mg LY2623091 First Then 10 mg LY2623091: Participants received 0.2 mg LY2623091 administered orally, QD for 21 days in treatment period 1 followed by a minimum 28-day washout period before receiving 10 mg LY2623091 for 21 days in treatment period 2. On Day 1 through Day 20, participants were in a fed state and on Day 21 participants were in a fasted state.
- 0.2 mg LY2623091 First Then 50 mg Eplerenone: Participants received 0.2 mg LY2623091 administered orally, QD for 21 days in treatment period 1 followed by a minimum 28-day washout period before receiving 50 mg Eplerenone for 21 days in treatment period 2. On Day 1 through Day 20, participants were in a fed state and on Day 21 participants were in a fasted state.
- 0.2 mg LY2623091 First Then 1.5 mg LY2623091: Participants received 0.2 mg LY2623091 administered orally, QD for 21 days in treatment period 1 followed by a minimum 28-day washout period before receiving 1.5 mg LY2623091 for 21 days in treatment period 2. On Day 1 through Day 20, participants were in a fed state and on Day 21 participants were in a fasted state.
- 10mg LY2623091 First Then 50mg Eplerenone: Participants received 10 mg LY2623091 administered orally, QD for 21 days in treatment period 1 followed by a minimum 28-day washout period before receiving 50 mg Eplerenone for 21 days in treatment period 2. On Day 1 through Day 20, participants were in a fed state and on Day 21 participants were in a fasted state.
- 10mg LY2623091 First Then 0.2 mg LY2623091: Participants received 10 mg LY2623091 administered orally, QD for 21 days in treatment period 1 followed by a minimum 28-day washout period before receiving 0.2 mg LY2623091 for 21 days in treatment period 2. On Day 1 through Day 20, participants were in a fed state and on Day 21 participants were in a fasted state.
- 10 mg LY2623091 First Then 1.5 mg LY2623091: Participants received 10 mg LY2623091 administered orally, QD for 21 days in treatment period 1 followed by a minimum 28-day washout period before receiving 1.5 mg LY2623091 for 21 days in treatment period 2. On Day 1 through Day 20, participants were in a fed state and on Day 21 participants were in a fasted state.
Period: Treatment Period 1 (21 Days)
Arm/Group | 1.5 mg LY2623091 First Then 10 mg LY2623091 | 1.5 mg LY2623091 First Then 50 mg Eplerenone | 1.5 mg LY2623091 First Then 0.2 mg LY2623091 | 50mg Eplerenone First Then 0.2 mg LY2623091 | 50mg Eplerenone First Then 1.5 mg LY2623091 | 50mg Eplerenone First Then 10 mg LY2623091 | 0.2 mg LY2623091 First Then 10 mg LY2623091 | 0.2 mg LY2623091 First Then 50 mg Eplerenone | 0.2 mg LY2623091 First Then 1.5 mg LY2623091 | 10mg LY2623091 First Then 50mg Eplerenone | 10mg LY2623091 First Then 0.2 mg LY2623091 | 10 mg LY2623091 First Then 1.5 mg LY2623091
Started | 3 | 4 | 4 | 3 | 4 | 3 | 3 | 5 | 3 | 3 | 3 | 4
Received at Least 1 Dose of Study Drug | 3 | 4 | 4 | 3 | 4 | 3 | 3 | 5 | 3 | 3 | 3 | 4
Completed | 3 | 4 | 4 | 3 | 4 | 3 | 3 | 4 | 3 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Washout (at Least 28 Days)
Arm/Group | 1.5 mg LY2623091 First Then 10 mg LY2623091 | 1.5 mg LY2623091 First Then 50 mg Eplerenone | 1.5 mg LY2623091 First Then 0.2 mg LY2623091 | 50mg Eplerenone First Then 0.2 mg LY2623091 | 50mg Eplerenone First Then 1.5 mg LY2623091 | 50mg Eplerenone First Then 10 mg LY2623091 | 0.2 mg LY2623091 First Then 10 mg LY2623091 | 0.2 mg LY2623091 First Then 50 mg Eplerenone | 0.2 mg LY2623091 First Then 1.5 mg LY2623091 | 10mg LY2623091 First Then 50mg Eplerenone | 10mg LY2623091 First Then 0.2 mg LY2623091 | 10 mg LY2623091 First Then 1.5 mg LY2623091
Started | 3 | 4 | 4 | 3 | 4 | 3 | 3 | 4 | 3 | 3 | 3 | 4
Completed | 3 | 4 | 4 | 3 | 4 | 1 | 3 | 4 | 3 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (21 Days)
Arm/Group | 1.5 mg LY2623091 First Then 10 mg LY2623091 | 1.5 mg LY2623091 First Then 50 mg Eplerenone | 1.5 mg LY2623091 First Then 0.2 mg LY2623091 | 50mg Eplerenone First Then 0.2 mg LY2623091 | 50mg Eplerenone First Then 1.5 mg LY2623091 | 50mg Eplerenone First Then 10 mg LY2623091 | 0.2 mg LY2623091 First Then 10 mg LY2623091 | 0.2 mg LY2623091 First Then 50 mg Eplerenone | 0.2 mg LY2623091 First Then 1.5 mg LY2623091 | 10mg LY2623091 First Then 50mg Eplerenone | 10mg LY2623091 First Then 0.2 mg LY2623091 | 10 mg LY2623091 First Then 1.5 mg LY2623091
Started | 3 | 4 | 4 | 3 | 4 | 1 | 3 | 4 | 3 | 3 | 3 | 4
Completed | 3 | 3 | 4 | 3 | 4 | 1 | 3 | 4 | 3 | 3 | 3 | 4
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1.5 mg LY2623091 First Then 10 mg LY2623091 | 1.5 mg LY2623091 First Then 50 mg Eplerenone | 1.5 mg LY2623091 First Then 0.2 mg LY2623091 | 50mg Eplerenone First Then 0.2 mg LY2623091 | 50mg Eplerenone First Then 1.5 mg LY2623091 | 50mg Eplerenone First Then 10 mg LY2623091 | 0.2 mg LY2623091 First Then 10 mg LY2623091 | 0.2 mg LY2623091 First Then 50 mg Eplerenone | 0.2 mg LY2623091 First Then 1.5 mg LY2623091 | 10mg LY2623091 First Then 50mg Eplerenone | 10mg LY2623091 First Then 0.2 mg LY2623091 | 10 mg LY2623091 First Then 1.5 mg LY2623091 | Total
Number analyzed (Participants) | 3 | 4 | 4 | 3 | 4 | 3 | 3 | 5 | 3 | 3 | 3 | 4 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 4 | 2 | 4 | 3 | 2 | 5 | 2 | 3 | 2 | 4 | 37
  >=65 years | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 0 | 2 | 2 | 1 | 3 | 2 | 0 | 1 | 2 | 17
  Male | 1 | 2 | 4 | 3 | 2 | 1 | 2 | 2 | 1 | 3 | 2 | 2 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 3 | 2 | 4 | 3 | 3 | 3 | 3 | 4 | 1 | 2 | 3 | 3 | 34
  Black/African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 4
  Mixed | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Bulgaria | 2 | 2 | 2 | 2 | 2 | 1 | 1 | 3 | 0 | 1 | 1 | 3 | 20
  South Africa | 1 | 2 | 1 | 1 | 2 | 2 | 2 | 2 | 3 | 2 | 2 | 1 | 21
  Macedonia | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 21 in Proteinuria Based on 24-hours Pooled Urine
Description: Proteinuria was the presence of excess serum protein in the urine. Proteinuria was calculated for each participant after each treatment period. Change was calculated as (Day 21 post-treatment value) minus (baseline value).
Time Frame: Over 24 hours at Baseline and on Day 21
Population: All participants who received any study drug and had proteinuria values. Participants were analyzed based on the treatment they received.
Measure: Mean (Standard Deviation); unit: milligrams/24 hours (mg/24 h)
Groups:
- 0.2 mg LY2623091: 0.2 mg LY2623091 capsules were administered to participants in either Period 1 or Period 2. In each period 0.2 mg LY2623091 was administered orally, QD for 21 days. On Day 1 through Day 20 participants were in a fed state and on Day 21 participants were in a fasted state. There was a minimum 28-day Washout Period between Period 1 and Period 2.
- 1.5 mg LY2623091: 1.5 mg LY2623091 capsules were administered to participants in either Period 1 or Period 2. In each period 1.5 mg LY2623091 was administered orally, QD for 21 days. On Day 1 through Day 20 participants were in a fed state and on Day 21 participants were in a fasted state. There was a minimum 28-day Washout Period between Period 1 and Period 2.
- 10 mg LY2623091: 10 mg LY2623091 capsules were administered to participants in either Period 1 or Period 2. In each period 10 mg LY2623091 was administered orally, QD for 21 days. On Day 1 through Day 20 participants were in a fed state and on Day 21 participants were in a fasted state. There was a minimum 28-day Washout Period between Period 1 and Period 2.
- 50 mg Eplerenone: 50 mg Eplerenone capsules were administered to participants in either Period 1 or Period 2. In each period 50 mg Eplerenone was administered orally, QD for 21 days. On Day 1 through Day 20 participants were in a fed state and on Day 21 participants were in a fasted state. There was a minimum 28-day Washout Period between Period 1 and Period 2.
Arm/Group | 0.2 mg LY2623091 | 1.5 mg LY2623091 | 10 mg LY2623091 | 50 mg Eplerenone
Number analyzed (Participants) | 20 | 22 | 17 | 21
milligrams/24 hours (mg/24 h) | -98.9 (1450.56) | -19.7 (876.85) | 119.4 (1923.11) | 273.7 (1280.34)

2. Secondary Outcome: Change From Baseline to Day 21 in Potassium Clearance Following an Oral Potassium Challenge
Description: Urine potassium clearance is defined as the amount of renal potassium excreted per volume of urine from participant's pooled urine. The oral potassium challenge consisted of 35 milliequivalents (mEq) potassium administered over 10 minutes as a flavored potassium chloride solution. Change was calculated as (Day 21 values) minus (baseline values).
Time Frame: Over 0-6 hours at Baseline and on Day 21
Population: All participants who received any study drug and had potassium clearance values. Participants were analyzed based on the treatment they received.
Measure: Mean (Standard Deviation); unit: Hour*millimoles per liter (h*mmol/L)
Arm/Group | 0.2 mg LY2623091 | 1.5 mg LY2623091 | 10 mg LY2623091 | 50 mg Eplerenone
Number analyzed (Participants) | 10 | 10 | 8 | 8
Hour*millimoles per liter (h*mmol/L) | 0.097 (0.263) | -0.122 (0.393) | -0.174 (0.243) | -0.019 (0.245)

3. Secondary Outcome: Pharmacokinetics (PK): Area Under the Plasma Concentration Time Curve During the Dosing Period of LY2623091 (AUC0-τ)
Time Frame: Predose, 1, 2, 4, 8, 12, and 24 hours postdose on Day 20 of Treatment Periods 1 and 2
Population: All participants who received LY2623091 and had AUC0-τ values. Participants were analyzed based on the treatment they received.
Measure: Mean (Standard Deviation); unit: hours*nanogram/milliliter (h*ng/mL)
Arm/Group | 0.2 mg LY2623091 | 1.5 mg LY2623091 | 10 mg LY2623091
Number analyzed (Participants) | 20 | 22 | 17
hours*nanogram/milliliter (h*ng/mL) | 75.321 (31.927) | 526.640 (177.834) | 3096.658 (1448.414)

4. Secondary Outcome: PK: Maximum Plasma Concentration (Cmax) of LY2623091
Time Frame: Predose, 1, 2, 4, 8, 12, and 24 hours postdose on Day 20 of Treatment Periods 1 and 2
Population: All participants who received LY2623091and had Cmax values. Participants were analyzed based on the treatment they received.
Measure: Mean (Standard Deviation); unit: nanograms/milliliter (ng/mL)
Arm/Group | 0.2 mg LY2623091 | 1.5 mg LY2623091 | 10 mg LY2623091
Number analyzed (Participants) | 20 | 22 | 17
nanograms/milliliter (ng/mL) | 4.540 (2.003) | 31.722 (10.325) | 187.441 (87.858)

5. Other Pre Specified Outcome: The Number of Participants Who Died While on Study
Time Frame: Baseline up to end of Treatment Period 2 plus 10-day follow-up (80 days)
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.2 mg LY2623091 | 1.5 mg LY2623091 | 10 mg LY2623091 | 50 mg Eplerenone
Number analyzed (Participants) | 21 | 22 | 17 | 21
Participants | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Description: Participants were randomized to 1 of 4 treatment arms, 3 LY2623091 (LY) and 1 Eplerenone (Epl). Each participated in 2 treatment periods and a washout period. Participants who received LY in Period 1 were randomized to a different LY arm or Epl arm in Period 2. Participants who received Epl in Period 1 were randomized to an LY arm in Period 2.
Groups:
- 0.2 mg LY2623091: 0.2 mg LY2623091 capsules were administered to participants in either Period 1 or Period 2. In each period 0.2 mg LY2623091 was administered orally, QD for 21 days, on Day 1 through Day 20 participants were in a fed state and on Day 21 participants were in a fasted state. Participants went through a minimum 28-day Washout Period between Period 1 and Period 2.
- 1.5 mg LY2623091: 1.5 mg LY2623091 capsules were administered to participants in either Period 1 or Period 2. In each period 1.5 mg LY2623091 was administered orally, QD for 21 days, on Day 1 through Day 20 participants were in a fed state and on Day 21 participants were in a fasted state. Participants went through a minimum 28-day Washout Period between Period 1 and Period 2.
- 10 mg LY2623091: 10 mg LY2623091 capsules were administered to participants in either Period 1 or Period 2. In each period 10 mg LY2623091 was administered orally, QD for 21 days, on Day 1 through Day 20 participants were in a fed state and on Day 21 participants were in a fasted state. Participants went through a minimum 28-day Washout Period between Period 1 and Period 2.
- 50 mg Eplerenone: 50 mg Eplerenone capsules were administered to participants in either Period 1 or Period 2. In each period 50 mg Eplerenone was administered orally, QD for 21 days, on Day 1 through Day 20 participants were in a fed state and on Day 21 participants were in a fasted state. Participants went through a minimum 28-day Washout Period between Period 1 and Period 2.
Arm/Group | 0.2 mg LY2623091 | 1.5 mg LY2623091 | 10 mg LY2623091 | 50 mg Eplerenone
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/22 | 0/17 | 1/21
Other Adverse Events (participants affected / at risk) | 9/21 | 8/22 | 8/17 | 10/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.2 mg LY2623091 (N=21) | 1.5 mg LY2623091 (N=22) | 10 mg LY2623091 (N=17) | 50 mg Eplerenone (N=21)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arterial insufficiency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.2 mg LY2623091 (N=21) | 1.5 mg LY2623091 (N=22) | 10 mg LY2623091 (N=17) | 50 mg Eplerenone (N=21)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lip blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dacryocystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arterial insufficiency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days